CLINICAL TRIAL: NCT06561711
Title: Optimization of Minocycline-containing Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Treatment: a Multicentre, Randomized Controlled Trial
Brief Title: Optimization of Minocycline for Helicobacter Pylori Rescue Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjhy20240816
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; rescue therapy; minocycline; tetracycline
MeSH Terms: conditions — cyclopia sequence | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Tetracycline; Metronidazole; Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Minocycline group A (Experimental): Vonoprazan 20mg bid, Bismuth Potassium Citrate 300mg qid, Minocycline 50mg tid, Metronidazole 400mg tid
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Minocycline,Metronidazole
- Minocycline group B (Experimental): Vonoprazan 20mg bid, Bismuth Potassium Citrate 300mg qid, Minocycline 50mg bid, Metronidazole 400mg qid
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Minocycline,Metronidazole
- Minocycline group C (Experimental): Vonoprazan 20mg bid, Bismuth Potassium Citrate 300mg qid, Minocycline 50mg bid, Metronidazole 400mg tid
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Minocycline,Metronidazole
- Tetracycline group (Active Comparator): Vonoprazan 20mg bid, Bismuth Potassium Citrate 300mg qid, Tetracycline 500mg qid, Metronidazole 400mg qid
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Tetracycline,Metronidazole

INTERVENTIONS:
Drug: Vonoprazan — Potassium competitive acid blocker
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Tetracycline,Metronidazole — Antibiotics for H. pylori eradication
  Arms: Tetracycline group
Drug: Minocycline,Metronidazole — Antibiotics for H. pylori eradication
  Arms: Minocycline group A; Minocycline group B; Minocycline group C

SUMMARY:
The efficacy of bismuth-containing quadruple therapy with minocycline and metronidazole was not inferior to classical bismuth quadruple therapy for refractory H. pylori infection, though also accompanied with high occurrence of adverse events (55.4%). Optimization of minocycline-based regimen to achieve high eradication rate with fewer adverse events is imperative. This study aimed to compare the efficacy and tolerability of a 14-day bismuth-containing quadruple rescue therapy with different dosage of minocycline and metronidazole compared to classical bismuth quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with previous treatment experience

Exclusion Criteria:

* subjects naive to H. pylori treatment,
* under 18 or over 80 years old
* history of gastrectomy
* pregnant or lactating women
* Previous history of tuberculosis
* Allergy to any of the study drugs
* severe systemic diseases or malignancy
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 8 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or severe" (causing considerable interference with daily activities). In addition, blood test were messured to access function of liver and kidney.
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Songjiang Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University school of Medicine, Hangzhou, Zhejiang